CLINICAL TRIAL: NCT01194115
Title: Use of 48 Hour Course of Antibiotics to Prevent Surgical Site Infection in Obese Patients Undergoing Cesarean Delivery
Acronym: SSI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Cincinnati (Other)
Responsible Party: Principal Investigator, Rose Maxwell, Ph.D., Director of Clinical Research, University of Cincinnati
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Surgical Site Infection C-Sect
Record Dates: First submitted 2010-09-01; First posted 2010-09-02 (Estimated); Last update posted 2011-11-11 (Estimated); Status verified 2011-11

CONDITIONS: Surgical Site Infection in Obese Women Undergoing C-section
Keywords: surgical site infection; obesity; pregnancy; cesarean section; cesarean delivery
MeSH Terms: conditions — Surgical Wound Infection; Obesity | interventions — Cephalexin; Metronidazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cephalexin and metronidazole (Experimental): 500 mg cephalexin per oral every 8 hours for total of 6 doses; 500 mg metronidazole per oral every 8 hours for total of 6 doses
  Interventions: Drug: cephalexin & metronidazole
- Placebo/standard of care (Placebo Comparator): Placebo pills per oral every 8 hours for total of 6 doses
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: cephalexin & metronidazole — cephalexin at 500 mg per oral every 8 hours for a total of 6 doses
  Other Names: Keflex & Flagyl
  Arms: Cephalexin and metronidazole
Drug: placebo — placebo representing standard of care
  Arms: Placebo/standard of care

SUMMARY:
The purpose of this study is to evaluate if preoperative antibiotics, followed by 48 hour course of broad spectrum antibiotics prevents wound infection complications in patients that are obese who undergo cesarean section. Standard antibiotic prophylaxis in all weight women undergoing cesarean section is cefazolin prior to skin incision. It is the hypothesis that a prolonged, 48 hour course of broad spectrum antibiotics that are suited to prevent growth of normal vaginal flora will decrease the rate of surgical site infection in obese patients that are at a greatly increased risk of postoperative infections complications.

DETAILED DESCRIPTION:
We propose the conduction of a prospective, randomized, double-blinded clinical trial to evaluate an alternative prophylactic regimen for the prevention of surgical site infection. This study is to be conducted by the Department of Obstetrics at University Hospital. The intervention being studied will be the continuation of cephalexin and metronidazole for 48 hours. The primary outcome measure will be the development of infectious morbidity, including wound infection and endometritis, in the postoperative period.

In order to most effectively and accurately analyze our primary and secondary research outcomes, the investigators will standardize our surgical operation techniques in all ways feasible. These recommendations will be in concordance with American College of Obstetrics and Gynecology recommendations, as those generally accepted in the medical literature. All patients will undergo surgery in the same small group of HEPA filtration and positive air pressure operating rooms. Appropriate limitations on number of surgeons and assistants scrubbed for surgery as well as general OR traffic will be enforced. Patients will undergo hair clipping of the incision site when appropriate. Chlorhexidine skin decontamination will be the standard surgical site preparation. An antimicrobial, adhesive drape will be used. Prior to skin incision, cefazolin will be administered.

All patients to be considered for recruitment to this study will be undergoing delivery at University Hospital. Patients with an elevated BMI > 30 kg/m2 who undergo cesarean section will be considered for randomization either prior to delivery or in the first 7 hours after delivery, to accommodate the need for the first dose of study medication or placebo 8 hours after surgery. Only patients who agree to inclusion after informed consent will be randomized per protocol.

ELIGIBILITY:
Inclusion Criteria:

* BMI > 30kg/m*2
* Delivery via cesarean section
* consent to participate
* age 13 or older

Exclusion Criteria:

* known immunodeficiency syndromes
* non-English speaking
* known allergy to cephalosporins or metronidazole

Min Age: 13 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 475 (Estimated)
Dates: Start 2010-09; Primary Completion 2012-09 (Estimated)

PRIMARY OUTCOMES:
Surgical site infection | 6weeks post partum

SECONDARY OUTCOMES:
Febrile morbidity; Urinary tract infection; Endometritis | 6 weeks post partum

CONTACTS AND LOCATIONS:
Overall Officials: Carri Warshak, MD, Principal Investigator — University of Cincinnati
Locations (1):
- The Univeristy Hospital, Cincinnati, Ohio, United States

REFERENCES:
- [Background] Hofmeyr GJ, Smaill FM. WITHDRAWAN. Antibiotic prophylaxis for cesarean section. Cochrane Database Syst Rev. 2010 Jan 20;2010(1):CD000933. doi: 10.1002/14651858.CD000933.pub2. PMID 20091509
- [Background] Meyer NL, Hosier KV, Scott K, Lipscomb GH. Cefazolin versus cefazolin plus metronidazole for antibiotic prophylaxis at cesarean section. South Med J. 2003 Oct;96(10):992-5. doi: 10.1097/01.SMJ.0000060570.51934.14. PMID 14570343
- [Background] Robinson HE, O'Connell CM, Joseph KS, McLeod NL. Maternal outcomes in pregnancies complicated by obesity. Obstet Gynecol. 2005 Dec;106(6):1357-64. doi: 10.1097/01.AOG.0000188387.88032.41. PMID 16319263
- [Background] Elyan A, Mahran M, el-Maraghy M, Abou-Seeda M. Prophylactic intravenous metronidazole in cesarean section. Chemioterapia. 1984 Feb;3(1):67-70. PMID 6535654
- [Background] Tita AT, Owen J, Stamm AM, Grimes A, Hauth JC, Andrews WW. Impact of extended-spectrum antibiotic prophylaxis on incidence of postcesarean surgical wound infection. Am J Obstet Gynecol. 2008 Sep;199(3):303.e1-3. doi: 10.1016/j.ajog.2008.06.068. PMID 18771992
- [Derived] Valent AM, DeArmond C, Houston JM, Reddy S, Masters HR, Gold A, Boldt M, DeFranco E, Evans AT, Warshak CR. Effect of Post-Cesarean Delivery Oral Cephalexin and Metronidazole on Surgical Site Infection Among Obese Women: A Randomized Clinical Trial. JAMA. 2017 Sep 19;318(11):1026-1034. doi: 10.1001/jama.2017.10567. PMID 28975304